CLINICAL TRIAL: NCT04491006
Title: A Randomized, Placebo-Controlled, Translational Study of ATH-1017 in Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: A Study of ATH-1017 in Mild to Moderate Alzheimer's Disease
Acronym: ACT-AD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Athira Pharma (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATH-1017-AD-0202; U1111-1255-9714 (Other: WHO (UTN)); 18PTC-R-589358 (Other Grant/Funding Number: Alzheimer's Association); 1R01AG068268-01 (NIH)
Record Dates: First submitted 2020-07-23; First posted 2020-07-29 (Actual); Results first posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-05

CONDITIONS: Alzheimer Disease; Dementia of Alzheimer Type
Keywords: Alzheimer's Disease; Cognition; Dementia; ATH-1017; Memory Loss
MeSH Terms: conditions — Alzheimer Disease; Dementia; Memory Disorders

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel-group study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Dose (Experimental): Daily subcutaneous (SC) injection of Low Dose ATH-1017
  Interventions: Drug: ATH-1017
- High Dose (Experimental): Daily subcutaneous (SC) injection of High Dose ATH-1017
  Interventions: Drug: ATH-1017
- Placebo (Placebo Comparator): Daily subcutaneous (SC) injection of Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ATH-1017 — Daily subcutaneous (SC) injection of ATH-1017 in a pre-filled syringe
  Arms: High Dose; Low Dose
Drug: Placebo — Daily subcutaneous (SC) injection of Placebo in a pre-filled syringe
  Arms: Placebo

SUMMARY:
This study is designed to evaluate treatment effects of ATH-1017 (fosgonimeton) in mild to moderate Alzheimer's subjects with a randomized treatment duration of 26-weeks.

DETAILED DESCRIPTION:
This study is designed to assess the correlation of the functional translational biomarker P300 latency and change in ADAS-Cog11 induced by ATH-1017 therapy, over 26-week randomized, double-blind treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Age 55 to 85 years
* Mild-to-moderate AD dementia subjects, MMSE 14-24, CDR 1 or 2 at Screening
* Clinical diagnosis of dementia, due probably to AD, by Revised National Institute on Aging-Alzheimer's Association criteria (McKhann, 2011)
* Reliable and capable support person/caregiver
* Treatment-free or receiving stable acetylcholinesterase inhibitor (AChEI) treatment, defined as:

  * Treatment-naïve, OR
  * Subjects are on a stable, approved dose of an AChEI (except for donepezil at 23 mg PO) for at least 3 months before Screening OR
  * Subjects who received an AChEI in the past and discontinued 4 weeks prior to Screening

Key Exclusion Criteria:

* History of significant neurologic disease, other than AD, that may affect cognition, or concurrent with the onset of dementia
* History of unexplained loss of consciousness, and epileptic fits (unless febrile)
* Subject has atypical variant presentation of AD, if known from medical history, particularly non-amnestic AD
* History of brain MRI scan indicative of any other significant abnormality
* Hearing test result considered unacceptable for auditory ERP P300 assessment
* Diagnosis of severe major depressive disorder even without psychotic features
* Significant suicide risk
* History within 2 years of Screening, or current diagnosis of psychosis
* Myocardial infarction or unstable angina within the last 6 months
* Clinically significant (in the judgment of the investigator) cardiac arrhythmia (including atrial fibrillation), cardiomyopathy, or cardiac conduction defect (note: pacemaker is acceptable)
* Subject has either hypertension (supine diastolic blood pressure > 95 mmHg), or symptomatic hypotension in the judgment of the investigator
* Clinically significant ECG abnormality at Screening
* Renal insufficiency (serum creatinine > 2.0 mg/dL)
* Hepatic impairment with alanine aminotransferase or aspartate aminotransferase > 2 times the upper limit of normal, or Child-Pugh class B and C
* Malignant tumor within 3 years before Screening
* Memantine in any form, combination or dosage within 4 weeks prior to Screening
* Donepezil at 23 mg PO
* The subject has received active amyloid or tau immunization (i.e., vaccination for Alzheimer's disease) at any time, or passive immunization (i.e., monoclonal antibodies for Alzheimer's disease) within 6 months of Screening

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (7):
  - Syrentis Clinical Research, Santa Ana, California
  - Premiere Research Institute, West Palm Beach, Florida
  - iResearch Atlanta, Decatur, Georgia
  - Neurological Associates of Albany, Albany, New York
  - Center for Cognitive Health, Portland, Oregon
  - Evergreen Health Research Program, Kirkland, Washington
  - University of Washington, Seattle, Washington
- Australia (6):
  - Central Coast Neurosciences Research, Central Coast, New South Wales
  - St Vincent's Centre for Applied Medical Research, Translational Research Centre, Darlinghurst, New South Wales
  - Hammondcare Greenwich Hospital, Greenwich, New South Wales
  - KaRa MINDS, Macquarie Park, New South Wales
  - HammondCare, Malvern, Victoria
  - Australian Alzheimer's Research Organization, Nedlands, Western Australia

REFERENCES:
- [Background] McKhann GM, Knopman DS, Chertkow H, Hyman BT, Jack CR Jr, Kawas CH, Klunk WE, Koroshetz WJ, Manly JJ, Mayeux R, Mohs RC, Morris JC, Rossor MN, Scheltens P, Carrillo MC, Thies B, Weintraub S, Phelps CH. The diagnosis of dementia due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):263-9. doi: 10.1016/j.jalz.2011.03.005. Epub 2011 Apr 21. PMID 21514250

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at a total of 6 centers in Australia and 8 centers in the United States (US).
Pre-assignment Details: This was a multicenter, randomized, double-blind, placebo-controlled, parallel-group, dose-ranging study comparing ATH-1017 40 milligrams per day (mg/day) and ATH-1017 70 mg/day with placebo in participants with a clinical diagnosis of mild to moderate Alzheimer's disease (AD).
Groups:
- Placebo: Participants were randomized to receive placebo via subcutaneous (SC) injection once-daily (QD) preferably during daytime. The first SC injection of study drug was performed at site under supervision. The participant should withhold study drug administration on the day of subsequent clinic visits; study drug administration was done on site under supervision of site staff at these visits. Clinic visits took place on Day 1 and thereafter at Weeks 2, 6, 12, 16, 20, and 26, with a safety follow-up visit scheduled 4 weeks after completion of the double-blind period at Week 30
- ATH-1017 40 Milligrams (mg): Participants were randomized to receive ATH-1017 40 mg via SC injection QD preferably during daytime. The first SC injection of study drug was performed at site under supervision. The participant should withhold study drug administration on the day of subsequent clinic visits; study drug administration was done on site under supervision of site staff at these visits. Clinic visits took place on Day 1 and thereafter at Weeks 2, 6, 12, 16, 20, and 26, with a safety follow-up visit scheduled 4 weeks after completion of the double-blind period at Week 30
- ATH-1017 70 mg: Participants were randomized to receive ATH-1017 70 mg via SC injection QD preferably during daytime. The first SC injection of study drug was performed at site under supervision. The participant should withhold study drug administration on the day of subsequent clinic visits; study drug administration was done on site under supervision of site staff at these visits. Clinic visits took place on Day 1 and thereafter at Weeks 2, 6, 12, 16, 20, and 26, with a safety follow-up visit scheduled 4 weeks after completion of the double-blind period at Week 30
Period: Overall Study
Arm/Group | Placebo | ATH-1017 40 Milligrams (mg) | ATH-1017 70 mg
Started | 24 | 27 | 26
Completed | 23 | 24 | 19
Not Completed | 1 | 3 | 7
Not completed — Adverse Event | 0 | 3 | 5
Not completed — Withdrawal by Subject | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety Population: included all randomized participants who received at least one dose of the study medication.
Groups:
- Placebo: Participants were randomized to receive placebo via subcutaneous (SC) injection QD preferably during daytime. The first SC injection of study drug was performed at site under supervision. The participant should withhold study drug administration on the day of subsequent clinic visits; study drug administration was done on site under supervision of site staff at these visits. Clinic visits took place on Day 1 and thereafter at Weeks 2, 6, 12, 16, 20, and 26, with a safety follow-up visit scheduled 4 weeks after completion of the double-blind period at Week 30
- ATH-1017 40 mg: Participants were randomized to receive ATH-1017 40 mg via SC injection QD preferably during daytime. The first SC injection of study drug was performed at site under supervision. The participant should withhold study drug administration on the day of subsequent clinic visits; study drug administration was done on site under supervision of site staff at these visits. Clinic visits took place on Day 1 and thereafter at Weeks 2, 6, 12, 16, 20, and 26, with a safety follow-up visit scheduled 4 weeks after completion of the double-blind period at Week 30
- Total: Total of all reporting groups
Arm/Group | Placebo | ATH-1017 40 mg | ATH-1017 70 mg | Total
Number analyzed (Participants) | 24 | 27 | 26 | 77
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.0 (8.03) | 70.6 (6.54) | 73.4 (7.26) | 71.4 (7.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 12 | 39
  Male | 12 | 12 | 14 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 0 | 3
  Not Hispanic or Latino | 21 | 27 | 26 | 74
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 4
  White | 22 | 25 | 24 | 71
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Event-related Potential (ERP) P300 Latency at Baseline
Description: ERP P300 was a method of recording brain activity elicited by external stimuli, for example (e.g.), an oddball auditory stimulus, particularly of working memory access. The participant had to perform a task related to auditory stimuli in order to assess the P300 component (latency). The stimulus consisted of an oddball paradigm with 2 sound stimuli. Stimuli were presented through headphones and auditory stimulation for P300 was assessed in a recording lasting up to 10 minutes. It was calculated as the average across the pre-dose values at Baseline visit. Baseline was defined as Day 1.
Time Frame: At Baseline (Day 1)
Population: Modified Intent-to-Treat (mITT) Population: included all randomized participants who took at least one dose of the study medication and who completed at least one ERP P300 Baseline assessment and/or one post-Baseline ERP P300 assessment.
Measure: Mean (Standard Deviation); unit: Milliseconds (ms)
Arm/Group | Placebo | ATH-1017 40 mg | ATH-1017 70 mg
Number analyzed (Participants) | 23 | 26 | 25
Milliseconds (ms) | 361.5 (32.23) | 382.3 (40.18) | 375.3 (35.77)

2. Secondary Outcome: Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog11) at Baseline
Description: The ADAS-Cog11 was designed to measure cognitive symptom change in participants with Alzheimer's Disease (AD) and consisted of 11 tasks. It was performed to evaluate the correlation of ERP P300 latency and cognition. The standard 11 items (and corresponding score range) were: word recall (0-10), commands (0-5), constructional praxis (0-5), naming objects and fingers (0-5), ideational praxis (0-5), orientation (0-8), word recognition (0-12), spoken language ability (0-5), comprehension of spoken language (0-5), word-finding difficulty (0-5), and remembering test instructions (0-5). The test included 7 performance items and 4 clinician-rated items. The ADAS-Cog11 total score was the sum of all 11 individual items, with a total score ranging from 0 (no impairment) to 70 (severe impairment). Higher scores indicated more severe cognitive impairment. Baseline was defined as Day 1.
Time Frame: At Baseline (Day 1)
Population: mITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | ATH-1017 40 mg | ATH-1017 70 mg
Number analyzed (Participants) | 23 | 25 | 25
Scores on a scale | 23.0 (7.96) | 22.4 (8.94) | 20.7 (7.18)

ADVERSE EVENTS:
Time Frame: Up to Week 30
Description: Safety population which included all randomized participants who received at least one dose of the study medication.
Arm/Group | Placebo | ATH-1017 40 mg | ATH-1017 70 mg
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/27 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/24 | 3/27 | 0/26
Other Adverse Events (participants affected / at risk) | 18/24 | 24/27 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=24) | ATH-1017 40 mg (N=27) | ATH-1017 70 mg (N=26)
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cholinergic syndrome (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=24) | ATH-1017 40 mg (N=27) | ATH-1017 70 mg (N=26)
Injection site reaction (General disorders) | 1 | 17 | 21
Injection site vesicles (General disorders) | 0 | 4 | 1
Injection site pain (General disorders) | 0 | 3 | 1
Injection site induration (General disorders) | 1 | 1 | 1
Injection site nodule (General disorders) | 0 | 0 | 3
Injection site bruising (General disorders) | 1 | 0 | 1
Injection site erythema (General disorders) | 0 | 2 | 0
Injection site paraesthesia (General disorders) | 0 | 1 | 1
Injection site pruritus (General disorders) | 0 | 1 | 1
Injection site mass (General disorders) | 0 | 1 | 0
Injection site oedema (General disorders) | 0 | 0 | 1
Injection site rash (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 4 | 1
Chest discomfort (General disorders) | 0 | 1 | 1
Chest pain (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 0
Flushing (General disorders) | 0 | 1 | 0
Hot flush (General disorders) | 1 | 0 | 0
Induration (General disorders) | 0 | 1 | 0
Adverse drug reaction (General disorders) | 0 | 0 | 1
Immediate post-injection reaction (General disorders) | 0 | 1 | 0
Application site pruritus (General disorders) | 0 | 1 | 0
Feeling abnormal (General disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 4 | 2
Dizziness (Nervous system disorders) | 2 | 2 | 3
Dizziness postural (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 3 | 1
Extensor plantar response (Nervous system disorders) | 0 | 1 | 0
Hyporeflexia (Nervous system disorders) | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 1
Dementia Alzheimer's type (Nervous system disorders) | 0 | 1 | 0
Cholinergic syndrome (Nervous system disorders) | 0 | 1 | 0
Dysdiadochokinesis (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Facial paralysis (Nervous system disorders) | 1 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 1
Parosmia (Nervous system disorders) | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 1 | 6 | 5
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 2
Neutrophilia (Blood and lymphatic system disorders) | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 3
Constipation (Gastrointestinal disorders) | 2 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 2
Wound secretion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 2
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 2 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 4 | 1
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 1
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1 | 0
Depressive symptom (Psychiatric disorders) | 0 | 0 | 1
Dysphemia (Psychiatric disorders) | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 1
Intraocular pressure increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Eosinophil count increased (Investigations) | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Blepharitis (Eye disorders) | 1 | 0 | 0
Amaurosis fugax (Eye disorders) | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 2 | 0
Genital paraesthesia (Reproductive system and breast disorders) | 0 | 1 | 0
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT04491006/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-02): https://cdn.clinicaltrials.gov/large-docs/06/NCT04491006/SAP_001.pdf